CLINICAL TRIAL: NCT00962351
Title: Metal Ion Release From an FDA Approved Metal-on-Metal Hip Replacement Implant: A Multi-Center, Randomized Clinical Trial
Brief Title: Metal Ion Release From an FDA-Approved Metal-on-Metal Total Hip Replacement Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: University of Western Ontario, Canada (Other); DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, C. Anderson Engh, Jr., MD, Orthopaedic Surgeon, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AORI2009-0100
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Non-inflammatory Degenerative Joint Disease
Keywords: total hip replacement; primary cementless total hip arthroplasty; metal ion; metal-on-metal
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metal-on-Polyethylene (Other)
  Interventions: Procedure: Total Hip Replacement
- Metal-on-Metal, 28mm femoral head (Other)
  Interventions: Procedure: Total Hip Replacement
- Metal-on-Metal, 36mm femoral head (Other)
  Interventions: Procedure: Total Hip Replacement

INTERVENTIONS:
Procedure: Total Hip Replacement

SUMMARY:
This is a multi-center, randomized study to compare blood and urine cobalt, chromium, and titanium ion levels of a metal-on-metal articular bearing coupled with two different head sizes to that of a conventional metal-on-polyethylene bearing.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cementless primary total hip replacement
* Receiving acetabular cup of 52mm or greater
* Preoperative level of function and pain same as for conventional hip replacement
* Likelihood of obtaining relief of pain and improved function
* Full skeletal maturity
* Ability to follow instructions
* Good general health
* Willing to return for follow-up evaluations
* X-ray evaluation confirming the presence of NIDJD
* Femoral and acetabular bone stock that is sufficient, regarding strength and shape, and suitable to receive the implants

Exclusion Criteria:

* Age less than 40 years or greater than 80 years at time of surgery
* Patients templated to receive an acetabular component smaller than 52mm in diameter
* Presence of a previous prosthetic hip replacement device in the hip joint to be operated
* Previous girdlestone procedure or surgical fusion of the hip to be operated
* Acute femoral neck fracture
* Above knee amputation of the contralateral and/or ipsilateral leg
* Patients with a diagnosis of inflammatory degenerative arthritis
* Skeletally immature
* Evidence of active infections that may spread to other areas of the body
* The presence of a highly communicable disease that may limit follow-up
* Presence of known active metastatic or neoplastic disease
* Significant neurologic or musculoskeletal disorders or disease that may adversely affect gait or weightbearing
* Any previous hip surgery or conditions that may interfere with the total hip replacement's survival or outcome
* Any patient believed to be unwilling or unable to comply with a rehabilitation program for a cementless total hip replacement or indicates difficulty to return for follow-up
* Patient is know to be pregnant, a prisoner, mentally incompetent, and/or alcohol or drug abuser
* Any patient who qualifies for inclusion in the study but refuses consent to participate in the study
* Any steroid therapy, local or systemic, within three months prior to surgery
* Patient requiring structural bone grafts in order to support the prosthetic components or to shape the bone to receive the implants
* Patient has known allergies to metal, e.g., jewelry
* Any patient not meeting all radiographic and clinical parameters for inclusion

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-10; Primary Completion 2010-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
cobalt, chromium, and titanium ion levels in blood and urine | Pre-op, 6 months, 1 year, 2 years, 3 years, 5 years

SECONDARY OUTCOMES:
Hip function | Pre-op, 6 months,1 year, 2 years, 3 years, 5 years
Durability | 6 months, 1 year, 2 years, 3 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: C. Anderson Engh, Jr., MD, Principal Investigator — Anderson Orthopaedic Research Institute; Steven J. MacDonald, MD, Principal Investigator — Department of Orthopaedic Surgery, University of Western Ontario
Locations (2):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States
- Department of Orthopaedic Surgery, University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Result] Engh CA Jr, MacDonald SJ, Sritulanondha S, Thompson A, Naudie D, Engh CA. 2008 John Charnley award: metal ion levels after metal-on-metal total hip arthroplasty: a randomized trial. Clin Orthop Relat Res. 2009 Jan;467(1):101-11. doi: 10.1007/s11999-008-0540-9. Epub 2008 Oct 15. PMID 18855089